CLINICAL TRIAL: NCT04443166
Title: The Synergistic Effects of Intra-articular Hyaluronic Acid and Platelet-rich Plasma Injections on Knee Osteoarthritis
Acronym: HAPRP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: N202002101
Record Dates: First submitted 2020-06-10; First posted 2020-06-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Osteoarthritis Knees Both

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group A (Experimental): At the beginning of the study (T0), group A will receive one course of PRP+HA program and group B will receive one HA course (a single HA injection (Hyajoint) weekly for 3 weeks). The PRP+HA program includes 3 HA injections and a single PRP injection (Arthrex double syringe system).
  Interventions: Combination Product: A platelet-rich plasma (PRP)+ hyaluronic acid (HA) program
- Group B (Active Comparator): In the 6th month, alternately, group B will receive one PRP+HA program and group A will receive one HA course.
  Interventions: Combination Product: A platelet-rich plasma (PRP)+ hyaluronic acid (HA) program

INTERVENTIONS:
Combination Product: A platelet-rich plasma (PRP)+ hyaluronic acid (HA) program — a combination of intra-articular knee injection with platelet-rich plasma (PRP) and hyaluronic acid (HA)
  Other Names: A hyaluronic acid (HA) course (a single HA injection (Hyajoint) weekly for 3 weeks)

SUMMARY:
Although intra-articular knee injection with platelet-rich plasma (PRP) may have better outcomes than using hyaluronic acid (HA) for people with knee osteoarthritis (OA), it is expensive to use PRP. Programs with a combination of PRP and HA (PRP+HA) showed good results in vitro and animal studies. This 2-year study aims to clarify the short- and long-term effectiveness of the PRP+HA program for knee OA.

The study will recruit 60 persons aged between 50 and 80 years who have experienced symptomatic knee OA for 6 months or more and have a radiographic picture of knee OA of grades 1-3, based on the Kellegren-Lawrence scale. Those who have diabetes, fever, anemia (Hb <10 g/dl), thrombocytopenia (platelet count <150000/ml), a blood-clotting disease, knee deformity (genu valgum/varum >20 degrees), impaired leg mobility secondary to neuromuscular diseases or a bony fracture, impaired mental function, severe cardiopulmonary impairment, taking anticoagulants long-term, a history of intra-articular steroid injection in the prior 1 year, a history of knee injury involving ligaments and menisci, and a history of malignancy are excluded.

All participants will be randomly divided into group A and group B. At the beginning of the study (T0), group A will receive one course of PRP+HA program and group B will receive one HA course (a single HA injection (Hyajoint) weekly for 3 weeks). The PRP+HA program includes 3 HA injections and a single PRP injection (Arthrex double syringe system). In the 6th month, alternately, group B will receive one PRP+HA program and group A will receive one HA course. The study has 3 outcome assessment tools including a self-administered Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Index, measurement of quadriceps strength with a digital handheld dynamometer, and measurement of femoral condylar cartilage thickness with musculoskeletal ultrasound. The investigators will conduct those assessments in the beginning (T0) of the study and the following 1st (T1), 3rd (T2), 6th (T3), and 9th (T4) months.

In the 18th month following the beginning of the study, both groups will receive a booster course of PRP+HA program. During the first week of the program, group A will receive a HA injection before the PRP injection and group B will receive the HA injection after the PRP injection. The investigators will conduct the long-term assessments in the 12th (T5), 15th (T6), 18th (T7), and 21st (T8) months since the beginning of the study.

DETAILED DESCRIPTION:
People aged >65 years are over 14% in Taiwan since the year 2018. Knee osteoarthritis (OA) is prevalent among elderly people. People with knee OA often have knee pain and stiffness as well as compromised their walking performance and quality of daily life. Although intra-articular knee injection with platelet-rich plasma (PRP) may have better outcomes than using hyaluronic acid (HA), it is expensive to use PRP. Programs with a combination of PRP and HA (PRP+HA) showed good results in vitro and animal studies. This 2-year study aims to clarify the short- and long-term effectiveness of the PRP+HA program for knee OA. The study will also assess the effectiveness of a booster course of PRP+HA program in the second year.

The study will recruit 60 persons aged between 50 and 80 years who have experienced symptomatic knee OA for 6 months or more and have a radiographic picture of knee OA of grades 1-3, based on the Kellegren-Lawrence scale. Those who have diabetes, fever, anemia (Hb <10 g/dl), thrombocytopenia (platelet count <150000/ml), a blood-clotting disease, knee deformity (genu valgum/varum >20 degrees), impaired leg mobility secondary to neuromuscular diseases or a bony fracture, impaired mental function who have difficulty in completing outcome assessments, severe cardiopulmonary impairment, taking anticoagulants long-term, a history of intra-articular steroid injection in the prior 1 year, a history of knee injury involving ligaments and menisci, and a history of malignancy are excluded.

All participants will be randomly divided into group A and group B. At the beginning of the study (T0), group A will receive one course of PRP+HA program and group B will receive one HA course (a single HA injection (Hyajoint) weekly for 3 weeks). The PRP+HA program includes 3 HA injections and a single PRP injection (Arthrex double syringe system). In the 6th month, alternately, group B will receive one PRP+HA program and group A will receive one HA course. The study has 3 outcome assessment tools including a self-administered Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Index, measurement of quadriceps strength with a digital handheld dynamometer, and measurement of femoral condylar cartilage thickness with musculoskeletal ultrasound. The investigators will conduct those assessments in the beginning (T0) of the study and the following 1st (T1), 3rd (T2), 6th (T3), and 9th (T4) months.

In the 18th month following the beginning of the study, both groups will receive a booster course of PRP+HA program. During the first week of the program, group A will receive a HA injection before the PRP injection and group B will receive the HA injection after the PRP injection. The investigators will conduct the long-term assessments in the 12th (T5), 15th (T6), 18th (T7), and 21st (T8) months since the beginning of the study.

ELIGIBILITY:
Inclusion Criteria:

* The study will recruit persons aged between 50 and 80 years who have experienced symptomatic knee OA for 6 months or more. They have a radiographic picture of knee OA of grades 1-3, based on the Kellegren-Lawrence scale.

Exclusion Criteria:

* Those who have diabetes, fever, anemia (Hb <10 g/dl), thrombocytopenia (platelet count <150000/ml), a blood-clotting disease, knee deformity (genu valgum/varum >20 degrees), impaired leg mobility secondary to neuromuscular diseases or a bony fracture, impaired mental function who have difficulty in completing outcome assessments, severe cardiopulmonary impairment, taking anticoagulants long-term, a history of intra-articular steroid injection in the prior 1 year, a history of knee injury involving ligaments and menisci, and a history of malignancy are excluded.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
changes in WOMAC index | in the beginning (T0) of the study and the following 1st (T1), 3rd (T2), 6th (T3), 9th (T4), 12th (T5), 15th (T6), 18th (T7), and 21st (T8) months.
  a self-administered Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Index
changes in quadriceps strength | in the beginning (T0) of the study and the following 1st (T1), 6th (T3), 12th (T5), 18th (T7), and 21st (T8) months.
  measurement of quadriceps strength with a digital handheld dynamometer
changes in cartilage thickness | in the beginning (T0) of the study and the following 1st (T1), 6th (T3), 12th (T5), 18th (T7), and 21st (T8) months.
  measurement of femoral condylar cartilage thickness with musculoskeletal ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Kwang-Hwa Chang, MD, Principal Investigator — Prof.

IPD SHARING:
Plan to Share IPD: No